CLINICAL TRIAL: NCT07113990
Title: Efficacy and Safety of Electroacupuncture Combined With rTMS on Motor Function Recovery After Stroke: A Multi-center Randomized Controlled Clinical Study
Brief Title: Electroacupuncture and rTMS for Post-Stroke Motor Recovery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jing Tao (Other)
Responsible Party: Sponsor-Investigator, Jing Tao, Professor, Fujian University of Traditional Chinese Medicine
Organization: Fujian University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FujianUTCM-7
Record Dates: First submitted 2025-08-03; First posted 2025-08-11 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Stroke
Keywords: Electroacupuncture; Repetitive Transcranial Magnetic Stimulation (rTMS); Stroke Rehabilitation; Motor Function ; Multicenter Randomized Controlled Trial
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active rTMS + Active EA group (Experimental)
  Interventions: Procedure: Active EA; Device: Active rTMS
- Active rTMS + Sham EA group (Sham Comparator)
  Interventions: Procedure: Sham EA; Device: Active rTMS

INTERVENTIONS:
Procedure: Active EA — Participants will receive electroacupuncture once daily for 2 consecutive weeks (total 10 sessions). Disposable sterile needles will be inserted at standardized acupoints to achieve de qi, then connected to an electroacupuncture device for 30 minutes per session.
  Arms: Active rTMS + Active EA group
Procedure: Sham EA — Participants will receive sham electroacupuncture once daily for 2 consecutive weeks (total 10 sessions). Disposable blunt needles will be placed at the same acupoints without skin penetration or electrical stimulation, with the electroacupuncture device turned on but delivering no current, for 30 minutes per session.
  Arms: Active rTMS + Sham EA group
Device: Active rTMS — Participants will receive high-frequency rTMS to the ipsilesional M1 area once daily for 2 consecutive weeks (total 10 sessions). Stimulation will be delivered with a MagPro R30 stimulator at 10 Hz, 1600 pulses per session, 4-second trains with 41-second inter-train intervals.

SUMMARY:
This study aims to evaluate the combined efficacy of repetitive Transcranial Magnetic Stimulation (rTMS) and Electroacupuncture (EA) in improving motor function recovery post-stroke, compared to rTMS combined with sham EA. Participants will receive either active EA or sham EA alongside standard rTMS treatment. Outcomes will be assessed using standardized clinical scales and neuroimaging techniques to explore underlying neuroplasticity mechanisms.

DETAILED DESCRIPTION:
Motor impairment is a major cause of disability following stroke, with central and peripheral neuromodulation strategies showing potential for functional recovery. Repetitive transcranial magnetic stimulation (rTMS) has been shown to promote neuroplasticity and enhance cortical excitability. Electroacupuncture (EA), by increasing somatosensory input, may further strengthen sensorimotor integration and cortical remodeling. However, limited clinical trials have systematically evaluated the synergistic effect of rTMS combined with EA.

This multi-center randomized controlled clinical study aims to assess the efficacy of combining rTMS and EA in improving motor function post-stroke. Outcome measures include clinical scales (FMA, ARAT, FAC), kinematic parameters, electrophysiological indices (EEG, EMG, TMS), blood biomarkers, and resting-state fMRI. The study is designed to explore central-peripheral neuroplasticity mechanisms and provide evidence for integrated rehabilitation approaches.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with stroke confirmed by neuroimaging (CT/MRI).
* First-ever stroke, unilateral hemispheric lesion, related to motor dysfunction.
* Age between 40 and 75 years.
* Duration from stroke onset between 2 weeks and 6 months.
* Brunnstrom stage II-IV.
* Right-handed.
* Able to understand instructions and voluntarily provide written informed consent.

Exclusion Criteria:

* History of epilepsy or familial epilepsy.
* Motor dysfunction due to non-vascular causes (e.g., tumor, trauma).
* Severe aphasia or cognitive impairment (MoCA < 18).
* Severe systemic complications (e.g., severe organ dysfunction, deep vein thrombosis).
* Presence of metallic implants or contraindications for MRI.
* Severe anxiety (HAMA > 7) or depression (HAMD > 8).
* Severe spasticity (modified Ashworth ≥ 2).
* Fear or intolerance of TMS or electroacupuncture.
* Pregnancy, breastfeeding, or concurrent participation in other clinical trials affecting outcomes.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment (FMA) | Baseline, 2 weeks post-intervention, 1month follow-up, 3months follow-up
  The Fugl-Meyer Assessment is used for rating motor function recovery after stroke. Scores range from 0 to 100, with higher scores indicating better motor performance.

SECONDARY OUTCOMES:
Arm Research Action Test (ARAT) | Baseline, 2 weeks post-intervention, 1month follow-up, 3months follow-up
  The Arm Research Action Test is used for assessing upper limb motor function across grasp, grip, pinch, and gross movement domains. Scores range from 0 to 57, with higher scores indicating better upper limb function.
Functional Ambulation Classification (FAC) | Baseline, 2 weeks post-intervention, 1month follow-up, 3months follow-up
  The Functional Ambulation Classification is used for evaluating the degree of ambulation independence. Scores range from 0 to 5, with higher scores indicating greater ambulation capability.
Modified Barthel Index (MBI) | Baseline, 2 weeks post-intervention, 1month follow-up, 3months follow-up
  The Modified Barthel Index is used for rating the level of independence in daily living activities. Scores range from 0 to 100, with higher scores indicating better functional independence.
Stroke-Specific Quality of Life Scale (SS-QOL) | Baseline, 2 weeks post-intervention, 1month follow-up, 3months follow-up
  The Stroke-Specific Quality of Life Scale is used for assessing health-related quality of life across 12 domains. Scores range from 49 to 245, with higher scores indicating better perceived quality of life.

OTHER OUTCOMES:
Kinematic Analysis of Upper Limb Motor Tasks | Baseline, 2 weeks post-intervention, 1month follow-up, 3months follow-up
  Optical motion capture of limb movement kinematics during functional tasks
Blood Biomarkers | Baseline, 2 weeks post-intervention
  Circulating neuroplasticity and inflammation biomarkers in venous blood samples.
Electrophysiological Assessments (EMG, EEG, TMS) | Baseline, 2 weeks post-intervention
  Electromyography (EMG), electroencephalography (EEG) and transcranial magnetic stimulation (TMS) assessments.
  Note: This outcome is planned to be conducted at selected sites depending on equipment availability and final coordination. The specific evaluation sites are under discussion.
fMRI | Baseline, 2 weeks post-intervention
  Structural and functional MRI acquired on a 3 T scanner. Note: This outcome will be assessed only at Fujian Provincial Hospital (Affiliated Hospital of Fuzhou University).

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Fuzhou University Affiliated Provincial Hospital, Fuzhou, Fujian
  - Fujian Provincial People's Hospital, Fuzhou, Fujian
  - Wenzhou Hospital of Traditional Chinese Medicine, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No